CLINICAL TRIAL: NCT03258554
Title: Randomized Phase II/III Trial of Radiotherapy With Concurrent MEDI4736 (Durvalumab) vs. Radiotherapy With Concurrent Cetuximab in Patients With Locoregionally Advanced Head and Neck Cancer With a Contraindication to Cisplatin
Brief Title: Radiation Therapy With Durvalumab or Cetuximab in Treating Patients With Locoregionally Advanced Head and Neck Cancer Who Cannot Take Cisplatin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01522; NCI-2017-01522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN004 (Other: NRG Oncology); NRG-HN004 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Squamous Cell Carcinoma of Unknown Primary; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Cetuximab; (225)Ac-DOTA-c(RGDyK); durvalumab; Immunoglobulin G; Disulfides; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cetuximab, radiation therapy) (Active Comparator): Patients receive cetuximab IV weekly over 60-120 minutes. Treatment repeats every week for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Beginning 5-7 days after first cetuximab dose, patients undergo IMRT 5 fractions per week for up to 7 weeks.
  Interventions: Biological: Cetuximab; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (durvalumab, radiation therapy) (Experimental): Patients receive durvalumab IV over 60 minutes every 4 weeks. Treatment repeats every 4 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Beginning week 2, patients undergo IMRT 5 fractions per week for up to 7 weeks.
  Interventions: Biological: Durvalumab; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm I (cetuximab, radiation therapy)
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Arm II (durvalumab, radiation therapy)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II/III trial studies how well radiation therapy works with durvalumab or cetuximab in treating patients with head and neck cancer that has spread to a local and/or regional area of the body who cannot take cisplatin. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cetuximab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. It is not known if radiation therapy with durvalumab will work better than the usual therapy of radiation therapy with cetuximab in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of radiotherapy (RT) with concurrent and adjuvant anti-PD-L1 therapy (MEDI4736 [durvalumab]) is safe in patients with locoregionally advanced head and neck cancer (HNC) who have a contraindication to cisplatin. (Lead-in) II. To test the hypothesis that concurrent RT and anti-PD-L1 therapy improves progression free survival (PFS) compared to standard therapy (RT with concurrent cetuximab) in patients with locoregionally advanced HNC who have a contraindication to cisplatin. (Phase II) III. To test the hypothesis that concurrent RT and anti-PD-L1 therapy improves overall survival compared to standard therapy (RT with concurrent cetuximab) in patients with locoregionally advanced HNC who have a contraindication to cisplatin. (Phase III)

SECONDARY OBJECTIVES:

I. To compare toxicity using Common Terminology Criteria for Adverse Events (CTCAE) and Patient Reported Outcomes (PRO)-CTCAE between patients treated with RT + anti-PD-L1 therapy versus RT/cetuximab.

II. To test the effect of anti-PD-L1 therapy in the subpopulation of patients with tumors that overexpress PD-L1.

III. To compare overall survival, response (at 4-month fludeoxyglucose F-18 [FDG]-positron emission tomography [PET]-computed tomography [CT]), locoregional failure, distant metastasis, and competing mortality in the two arms by known risk factors, including p16 status and omega score.

IV. To test the hypothesis that MEDI4736 (durvalumab) therapy arm will have less decline in the physical function domain of European Organization for Research and Treatment of Cancer Core Questionnaire (EORTC QLQ-C30 version 3.0) based on the change in score from baseline to 12 months from end of RT, compared to the cetuximab-RT arm in patients with locoregionally advanced HNC who have a contraindication to cisplatin.

V. To test the hypothesis that MEDI4736 (durvalumab) therapy arm at 1 year (from end of RT) will have less decline in swallowing related quality of life (QOL) using the M. D. Anderson Dysphagia Inventory (MDADI) total composite score, based on the change in score from baseline to 12 months from end of RT, compared to the cetuximab-RT arm in patients who are medically unfit for cisplatin.

VI. To compare swallowing related performance and function short and long term using the Performance Status Scale for Head & Neck Cancer Patients (PSS-HN).

VII. To evaluate gastrostomy tube retention rates between arms.

EXPLORATORY OBJECTIVES:

I. To test the hypothesis that radiation combined with MEDI4736 (durvalumab) enhances the adaptive immune response using three types of immunophenotyping compared to radiation combined with cetuximab.

II. To compare overall QOL short term (end RT-8 months) and long term (12-24 months from end of RT) between arms using the EORTC QLQ-C30 version 3.0/HN35.

III. To evaluate swallowing related QOL short term (end RT-8 months) and long term (12-24 months from end of RT) using the EORTC Head and Neck (HN)35 swallowing domain and MDADI (subscales) between arms in patients with locoregionally advanced HNC who have a contraindication to cisplatin.

IV. To evaluate patient reported fatigue using the fatigue items in the EORTC QLQ and PRO-CTCAE.

V. To compare clinician and patient reported toxicity using CTCAE and PRO CTCAE.

VI. To explore health utilities between cetuximab and MEDI4736 (durvalumab) RT using the European Quality of Life 5 Dimensional-5 Level (EQ5D-5L).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cetuximab intravenously (IV) weekly over 60-120 minutes. Treatment repeats every week for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Beginning 5-7 days after first cetuximab dose, patients undergo intensity modulated radiation therapy (IMRT) 5 fractions per week for up to 7 weeks.

ARM II: Patients receive durvalumab IV over 60 minutes every 4 weeks. Treatment repeats every 4 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Beginning week 2, patients undergo IMRT 5 fractions per week for up to 7 weeks.

After completion of study treatment, patients are followed up at 1 month, every 4 months for 1 year, every 6 months for 2 years, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION INCLUSION CRITERIA
* Patients must have pathologically confirmed, previously untreated, unresected squamous cell carcinoma of the larynx, hypopharynx, oropharynx, oral cavity, or carcinoma of unknown head/neck primary prior to step 1 registration; submission of hematoxylin and eosin (H&E) stained slides and formalin-fixed and paraffin-embedded (FFPE) tissue block (or punch biopsy of FFPE block) to the biospecimen bank at University of California, San Francisco (UCSF) for central review for oropharyngeal and unknown primaries and for p16 analysis for all other non-oropharyngeal primaries is mandatory for all patients; investigators should check with their pathology department regarding release of biospecimens before approaching patients about participation in the trial; for oropharyngeal and unknown primaries, submission of H&E and p16 stained slides (with the required block for PD-L1) to the biospecimen bank at UCSF for central review is also required prior to step 2 registration

  * Note: fine needle aspirates (FNA) samples are not acceptable since they do not provide enough material for PD-L1 and p16 testing; however, if a cell block derived from the FNA is available, it is allowable if there are sufficient cells present in the block for PD-L1 testing; Dr. Jordan will determine this upon receipt; for sites submitting FNA cell blocks for ALL patients they must do so within 7-10 business days from registering the patient; sites must confirm with their cytology/pathology labs to make sure they can provide the required material as the bank must be able to retain these samples for the mandatory testing
* Patients must have locoregionally advanced head and neck squamous cell carcinoma (HNSCC)

  * For p16-positive oropharyngeal/unknown primaries, American Joint Committee on Cancer [AJCC] 8th edition stage III and selected stage I-II based on smoking status in pack-years
  * For laryngeal, hypopharyngeal, and oral cavity primaries and p16-negative oropharyngeal/unknown primaries, AJCC 8th edition stage III-IVB
  * Based on the following minimum diagnostic workup within 60 days prior to step 1 registration:

    * General history and physical examination by a radiation oncologist or medical oncologist or ear, nose and throat (ENT) or head & neck surgeon
    * For larynx, hypopharynx, and base of tongue primaries, a laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) is required, unless the patient cannot tolerate or refuses
  * Imaging of the head and neck with a neck CT or magnetic resonance imaging (MRI) (with contrast, unless contraindicated) or PET/CT; note that the CT portion of the PET/CT must be of diagnostic quality, including contrast administration unless contraindicated. If the CT portion of the PET/CT study is low-dose (non-diagnostic), then an additional CT or MRI study with contrast (unless contraindicated) is required
  * Chest imaging: chest CT with and without contrast (unless contraindicated) or PET/CT
* Patients must have a contraindication to cisplatin as defined in the following bullet points; sites must complete the online tool at comogram.org prior to step 1 registration to determine if the patient is eligible; the scores must be recorded on a case report form (CRF)

  * Age >= 70 with moderate to severe comorbidity or vulnerability to cisplatin, defined as having one or more of the following conditions within 30 days prior to step 1 registration:

    * Modified Charlson Comorbidity Index >= 1
    * Adult Comorbidity Evaluation (ACE)-27 Index >= 1
    * Generalized Competing Event Model for Cancer Risk (GCE) omega PFS score < 0.80
    * Geriatric screening (G-8) score =< 14
    * Cancer and Aging Research Group (CARG) toxicity score >= 30%
    * Cumulative Illness Rating scale for Geriatrics (CIRS-G) score >= 4 OR
  * Age < 70 with severe comorbidity or vulnerability to cisplatin, defined as having two or more of the following conditions within 30 days prior to step 1 registration

    * Modified Charlson Comorbidity Index >= 1
    * ACE-27 Index >= 1
    * GCE omega PFS-score < 0.80
    * G-8 score =< 14
    * CARG Toxicity score >= 30%
    * CIRS-G score >= 4 OR
  * Age >= 18 with an absolute or relative contraindication to cisplatin, defined as one or more of the following within 30 days prior to step 1 registration:

    * Creatinine clearance (CC) > 30 and < 60 cc/min; for this calculation, use the Cockcroft-Gault formula
    * Zubrod performance status 2 prior to step 1 registration
    * Pre-existing peripheral neuropathy grade >= 1
    * History of hearing loss, defined as either:

      * Existing need of a hearing aid OR
      * >= 25 decibel shift over 2 contiguous frequencies on a pretreatment hearing test as clinically indicated
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 (within 14 days prior to step 1 registration)
* Platelets >= 100,000 cells/mm^3 (within 14 days prior to step 1 registration)
* Hemoglobin >= 9.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dl is acceptable) (within 14 days prior to step 1 registration)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 times institutional upper limit of normal (within 14 days prior to step 1 registration)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (within 14 days prior to step 1 registration)
* Measured creatinine clearance (CL) > 30 mL/min or calculated creatinine CL > 30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (within 14 days prior to step 1 registration)
* For women of childbearing potential, a negative serum or urine pregnancy test within 14 days prior to step 1 registration; Note: women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause; the following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* The patient or a legally authorized representative must provide study-specific informed consent prior to step 1 registration
* PRIOR TO STEP 2 REGISTRATION INCLUSION CRITERIA
* For patients with oropharyngeal or unknown primaries: p16 determination by immunohistochemistry (defined as greater than 70% strong nuclear or nuclear and cytoplasmic staining of tumor cells), confirmed by central pathology review

  * Note: for patients with oral cavity, laryngeal, and hypopharyngeal primaries, analysis of p16 status prior to step 2 registration/randomization is not required (p16 status will be analyzed centrally post-hoc); step 2 registration for these patients can be completed after step 1 registration

Exclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION EXCLUSION CRITERIA
* Prior invasive malignancy within the past 3 years (except for non-melanomatous skin cancer, and early stage treated prostate cancer); synchronous head and neck primaries are ineligible
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields

  * Note: Prior external beam radiotherapy is excluded, but iodine 131 is allowed
* Prior immunotherapy
* Prior systemic therapy, including cytotoxic chemotherapy, biologic/targeted therapy, or immune therapy for the study cancer
* Major surgery within 28 days prior to step 1 registration
* Proven evidence of distant metastases
* If both of the following conditions are present, the patient is ineligible:

  * =< 10 pack-year smoking history
  * p16-positive carcinoma of the oropharynx or unknown primary that are T0-3, N0-1 (AJCC 8th Edition)

    * Note: in the event that a registered patient with =< 10 pack-years has a p16-positive result on central review with the tumor and nodal stage T0-3, N0-1 (AJCC 8th Edition), then the site will be notified that the patient is ineligible
* Zubrod performance status >= 3
* Body weight =< 30 kg
* Patients with oral cavity cancer are excluded from participation if the patient is medically operable and resection of the primary tumor is considered technically feasible by an oral or head and neck cancers surgical subspecialist;(please consult the surgical oncology co-principal investigator [PI], Steven Chang, Doctor of Medicine [MD], if clarification is needed on an individual case)
* Sodium < 130 mmol/L or > 155 mmol/L (within 14 days of step 1 registration, unless corrected prior to step 1 registration)
* Potassium < 3.5 mmol/L or > 6 mmol/L (within 14 days of step 1 registration, unless corrected prior to step 1 registration)
* Fasting glucose < 40 mg/dl or > 400 mg/dl (within 14 days of step 1 registration, unless corrected prior to step 1 registration)
* Serum calcium (ionized or adjusted for albumin) < 7 mg/dl or > 12.5 mg/dl (within 14 days of step 1 registration, unless corrected prior to step 1 registration)
* Magnesium < 0.9 mg/dl or > 3 mg/dl (within 14 days of step 1 registration, unless corrected prior to step 1 registration)
* Unstable angina and/or congestive heart failure requiring hospitalization within 3 months prior to step 1 registration
* Transmural myocardial infarction within 3 months prior to step 1 registration
* Respiratory illness requiring hospitalization at the time of step 1 registration

  * Note: if the respiratory illness is resolved and the patient meets the eligibility status above, then the patient can be considered for the trial
* Idiopathic pulmonary fibrosis or other severe interstitial lung disease that requires oxygen therapy or is thought to require oxygen therapy within 1 year prior to step 1 registration
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Clinically apparent jaundice and/or known coagulation defects
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.)

  * The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia;
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement;
    * Any chronic skin condition that does not require systemic therapy;
    * Patients without active disease in the last 5 years may be included but only after consultation with the medical oncology study chair;
    * Patients with celiac disease controlled by diet alone
* History of active primary immunodeficiency including, but not limited to acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; Note: human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatment involved in this protocol may be immunosuppressive; patients with known HIV, CD4 counts >= 200/uL, and undetectable viral loads who are stable on an antiretroviral regimen may be included
* Current or prior use of immunosuppressive medication within 14 days before step 1 registration, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Receipt of live attenuated vaccination within 30 days prior to step 1 registration
* Medical or psychiatric illness which would compromise the patient's ability to tolerate treatment or limit compliance with study requirements
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for 6 months after the last dose of cetuximab or MEDI14736 (durvalumab); this exclusion is necessary because the treatment involved in this study may be significantly teratogenic; women who are breastfeeding are also excluded
* Prior allergic reaction or hypersensitivity to cetuximab or MEDI4736 (durvalumab) or any of study drug excipients
* History of allogenic organ transplantation
* Uncontrolled hypertension
* Uncontrolled cardiac arrhythmia
* Uncontrolled serious chronic gastrointestinal condition associated with diarrhea
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C; patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible; patients positive for hepatitis C (hepatitis C virus [HCV]) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren K Mell, Principal Investigator — NRG Oncology
Locations (256):
- United States (252):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Good Samaritan Hospital, Corvallis, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
- Canada (4):
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Derived] Mell LK, Torres-Saavedra PA, Wong SJ, Kish JA, Chang SS, Jordan RC, Liu T, Truong MT, Winquist EW, Takiar V, Wise-Draper T, Robbins JR, Rodriguez CP, Awan MJ, Beadle BM, Henson C, Narayan S, Spencer SA, Powell S, Dunlap N, Sacco AG, Hu KS, Park HS, Bauman JE, Harris J, Yom SS, Le QT. Radiotherapy with cetuximab or durvalumab for locoregionally advanced head and neck cancer in patients with a contraindication to cisplatin (NRG-HN004): an open-label, multicentre, parallel-group, randomised, phase 2/3 trial. Lancet Oncol. 2024 Dec;25(12):1576-1588. doi: 10.1016/S1470-2045(24)00507-2. Epub 2024 Nov 14. PMID 39551064
- See also: "Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive." — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were first registered for screening. Central pathology review confirmation of p16 determination was an enrollment requirement for participants with oropharyngeal or unknown primary tumors. Overall,196 of 200 screened participants were enrolled.
Groups:
- (Lead-in) RT + Durvalumab: Intensity-modulated radiation therapy (IMRT) for seven weeks, 5 fractions/week. Durvalumab 1500 mg IV starts two weeks prior to RT and continues every 4 weeks for a total of seven cycles in the absence of disease progression or unacceptable toxicity.
- RT + Cetuximab: IMRT for seven weeks, 5 fractions/week. Cetuximab 400 mg/m^2 IV starts one week prior to RT, then 250 mg/m^2 weekly for seven additional cycles in the absence of disease progression or unacceptable toxicity.
- RT + Durvalumab: IMRT for seven weeks, 5 fractions/week. Durvalumab 1500 mg IV starts two weeks prior to RT and continues every 4 weeks for a total of seven cycles in the absence of disease progression or unacceptable toxicity.
Period: Lead-in Component
Arm/Group | (Lead-in) RT + Durvalumab | RT + Cetuximab | RT + Durvalumab
Started | 10 | 0 | 0
Started Treatment | 10 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Randomized Component
Arm/Group | (Lead-in) RT + Durvalumab | RT + Cetuximab | RT + Durvalumab
Started | 0 | 63 | 123
Started Treatment | 0 | 61 | 119
Completed | 0 | 63 | 123
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants (i.e. for phase II, randomized)
Groups:
- (Lead-in) RT + Durvalumab; RT + Durvalumab: IMRT for seven weeks, 5 fractions/week. Durvalumab 1500 mg IV starts two weeks prior to RT and continues every 4 weeks for a total of seven cycles in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | (Lead-in) RT + Durvalumab | RT + Cetuximab | RT + Durvalumab | Total
Number analyzed (Participants) | 10 | 63 | 123 | 196
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 1 | 1 | 2 | 4
  50 - 59 years | 0 | 9 | 10 | 19
  60 - 69 years | 6 | 20 | 35 | 61
  70 - 79 years | 3 | 25 | 60 | 88
  ≥ 80 years | 0 | 8 | 16 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 9 | 21 | 31
  Male | 9 | 54 | 102 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 3 | 1 | 14
  Not Hispanic or Latino | 0 | 56 | 117 | 173
  Unknown or Not Reported | 0 | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 6 | 11 | 17
  White | 10 | 50 | 105 | 165
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 4 | 3 | 7
Zubrod performance status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 4 | 28 | 48 | 80
    1 | 6 | 27 | 60 | 93
    2 | 0 | 8 | 15 | 23
Modified Charlson Comorbidity Index (CCI) [Count of Participants; unit: Participants] — An assessment tool used to predict the mortality for a patient who may have a range of concurrent conditions (comorbidities). The score ranges from 0 (no comorbidities) to 35 (highest possible comorbidity load / highest risk of death). For this study, the CCI was modified to exclude the cancer questions: "Has the patient had cancer (other than basal cell skin cancer)?" and "Has the patient had a metastatic solid tumor?".
  Participants
    0 (no comorbidities) | 4 | 24 | 43 | 71
    ≥ 1 | 6 | 39 | 80 | 125
Primary tumor site and p16 status [Count of Participants; unit: Participants] — The biomarker p16 is used as a surrogate marker for human papillomavirus (HPV) infections and is a known prognostic factor in some head and neck cancers.
  Participants
    Oropharynx, p16-positive | 6 | 27 | 55 | 88
    Unknown, p16-positive | 0 | 3 | 3 | 6
    Oropharynx, p16-negative | 2 | 3 | 15 | 20
    Unknown, p16-negative | 0 | 0 | 1 | 1
    Oral cavity | 0 | 4 | 6 | 10
    Hypopharynx | 0 | 8 | 13 | 21
    Larynx | 2 | 18 | 30 | 50
T stage, clinical (AJCC 8) [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b. Lead-in component used 7th edition of AJCC; phase II component used 8th edition.
  Participants
    T0 | 0 | 3 | 4 | 7
    T1 | 3 | 7 | 11 | 21
    T2 | 2 | 16 | 38 | 56
    T3 | 3 | 20 | 42 | 65
    T4 | 2 | 11 | 15 | 28
    T4a | 0 | 6 | 11 | 17
    T4b | 0 | 0 | 2 | 2
N stage, clinical (AJCC 8) [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 7th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. The higher the number after the N, the greater the involvement of regional lymph nodes. Lead-in component used 7th edition of AJCC; phase II component used 8th edition.
  Participants
    N0 | 0 | 14 | 17 | 31
    N1 | 2 | 28 | 36 | 66
    N2 | 0 | 8 | 21 | 29
    N2a | 0 | 0 | 2 | 2
    N2b | 4 | 3 | 21 | 28
    N2c | 4 | 9 | 17 | 30
    N3 | 0 | 0 | 4 | 4
    N3a | 0 | 0 | 2 | 2
    N3b | 0 | 1 | 3 | 4
Smoking history: pack-years [Count of Participants; unit: Participants] — A way to measure the amount a person has smoked over a long period of time. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  Participants
    ≤ 10 pack-years | 4 | 21 | 35 | 60
    > 10 pack-years | 6 | 42 | 88 | 136
Comorbidity group [Count of Participants; unit: Participants]
  Absolute or relative contraindication to cisplatin | 6 | 52 | 104 | 162
  Age ≥ 70 with moderate to severe comorbidity or vulnerability to cisplatin | 1 | 4 | 12 | 17
  Age < 70 with severe comorbidity or vulnerability to cisplatin | 3 | 7 | 7 | 17
Number of comorbidity conditions [Count of Participants; unit: Participants]
  1 | 0 | 0 | 1 | 1
  2 | 1 | 3 | 5 | 9
  3 | 3 | 7 | 10 | 20
  4 | 0 | 14 | 23 | 37
  5 | 2 | 17 | 31 | 50
  ≥ 6 | 4 | 22 | 53 | 79
Stratification factor: Zubrod and modified CCI [Count of Participants; unit: Participants]
  Zubrod 0 and modified CCI 0 | NA — The lead-in component was not randomized and therefore participants were not stratified. | 13 | 20 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Zubrod 1-2 and/or modified CCI > 0 | NA — The lead-in component was not randomized and therefore participants were not stratified. | 50 | 103 | NA — Total not calculated because data are not available (NA) in one or more arms.
Stratification factor: primary site and p16 status [Count of Participants; unit: Participants]
  p16-positive oropharynx or unknown primary | NA — The lead-in component was not randomized and therefore participants were not stratified. | 30 | 58 | NA — Total not calculated because data are not available (NA) in one or more arms.
  p16-negative oropharynx or unknown primary, larynx, hypopharynx or oral cavity | NA — The lead-in component was not randomized and therefore participants were not stratified. | 33 | 65 | NA — Total not calculated because data are not available (NA) in one or more arms.
Stratification factor: T and N stage [Count of Participants; unit: Participants]
  T0-3 and N0-2 | NA — The lead-in component was not randomized and therefore participants were not stratified. | 45 | 88 | NA — Total not calculated because data are not available (NA) in one or more arms.
  T4 and/or N3 | NA — The lead-in component was not randomized and therefore participants were not stratified. | 18 | 35 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT) [Lead-in Phase]
Description: DLTs were collected to verify the safety of durvalumab with RT in this population. Safety was determined if ≤ 2 of 8 participants in the cohort had any DLT, in which case the study would proceed to phase II with that dose schedule (DS). The probability for the DS to be deemed too toxic, given a true toxicity rate ≥ 45%, is at least 78%. With a true toxicity rate ≤ 20%, the probability for the DS do be deemed safe is 80%. The full DLT definition does not fit here, but includes all grade 5 AEs, grade 3 or 4 AEs definitely or probably related to durvalumab (DPRD) except for specified AEs and situations, and incomplete or > 2-week delay completing RT due to immune toxicity DPRD. AEs were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, which grade severity from 1=mild to 5=death. Two alternate DSs with a delayed 2nd dose (to reduce/avoid doses concurrent with RT) would be tried if the initial DS was too toxic.
Time Frame: From start of durvalumab to 4 weeks after radiation therapy, approximately 13 weeks. Weekly during RT, at RT end, prior to adjuvant durvalumab, one month after end of RT.
Population: The first eight DLT evaluable participants in a given dose schedule cohort. An evaluable participant is defined as a participant who either (1) experienced a DLT and received at least one dose of durvalumab, or (2) received at least one dose of durvalumab and one fraction of radiation therapy (RT) and completed the DLT observation period (4 weeks after RT).
Measure: Count of Participants; unit: Participants
Arm/Group | (Lead-in) RT + Durvalumab
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Progression-free Survival (Percentage of Participants Alive Without Progression) [Phase II Primary]
Description: Progression (failure) is defined as local, regional, or distant disease progression, or death from any cause. Progression was assessed by imaging, clinical assessment, or biopsy.
  Failure time is defined as time from randomization to failure or last follow-up (censored). Failure rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided. Analysis was planned to occur after 69 failure events had been reported.
Time Frame: From randomization to last follow-up: weekly during RT, after end of RT: every 4 months for 1 year, every 6 months for 2 years, then annually. Additionally, every 4 weeks during adjuvant durvalumab. Maximum follow-up at time of analysis was 4.2 years.
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 63 | 123
percentage of participants | 63.7 [51.3 to 76.1] | 50.6 [41.5 to 59.8]
Statistical Analysis 1: Comparison: RT + Cetuximab vs RT + Durvalumab; Sixty-nine progression-free survival (PFS) events provides 0.80 power for a log-rank test with one-sided alpha of 0.20 to detect an improvement in PFS corresponding to a median of 2.35 years (RT+Durvalumab) compared to 1.53 years (RT+Cetuximab). A hazard ratio (RT+Durvalumab/RT+Cetuximab) ≤ 0.806 would indicate a rejection of the null hypothesis (no difference between the arms) and the study would continue to phase III; otherwise, the study would not continue to phase III; Test type: Superiority; p = 0.8878, Log Rank — One-sided significance level = 0.2; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.84 to 2.12] — Reference arm = radiation therapy + cetuximab

3. Primary Outcome: Overall Survival (Percentage of Participants Alive) [Originally Phase III Primary / Now Phase II Secondary]
Description: Overall survival (OS) time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided.
Time Frame: as for outcome 2
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RT+ Cetuximab: IMRT for seven weeks, 5 fractions/week. Cetuximab 400 mg/m^2 IV starts one week prior to RT, then 250 mg/m^2 weekly for seven additional cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | RT+ Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 63 | 123
percentage of participants | 77.5 [66.7 to 88.3] | 69.3 [60.8 to 77.8]
Statistical Analysis 1: Comparison: RT+ Cetuximab vs RT + Durvalumab; Test type: Superiority; p = 0.8175, Log Rank — One-side significance level = 0.025; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.74 to 2.28]

4. Secondary Outcome: Locoregional Failure (Percentage of Participants With Locoregional Failure)
Description: Locoregional progression is defined as local or regional progression or recurrence, death due to study cancer or unknown causes without documented progression. Progression was assessed by imaging, clinical assessment, or biopsy. Failure time is defined as time from randomization to failure, distant metastasis (competing risk), deaths from other causes (competing risk), or last follow-up (censored). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided.
Time Frame: as for outcome 2
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT+ Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 63 | 123
percentage of participants | 18.9 [10.0 to 29.9] | 31.3 [23.0 to 40.0]
Statistical Analysis 1: Comparison: RT+ Cetuximab vs RT + Durvalumab; Test type: Superiority; p = 0.1001, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.71, 95% CI 2-sided [0.89 to 3.28] — Reference level = RT+ Cetuximab

5. Secondary Outcome: Distant Metastasis (Percentage of Participants With Distant Metastasis)
Description: Failure is defined as the occurrence of distant metastasis. Failure time is defined as time from randomization to first occurrence of distant metastasis, local or regional progression or recurrence (competing risk), death (competing risk), or last follow-up (censored). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided.
Time Frame: as for outcome 2
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT+ Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 63 | 123
percentage of participants | 12.1 [5.3 to 22.0] | 9.5 [5.0 to 15.7]
Statistical Analysis 1: Comparison: RT+ Cetuximab vs RT + Durvalumab; Test type: Superiority; p = 0.5197, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.32 to 1.77] — Reference level = RT+ Cetuximab

6. Secondary Outcome: Competing Mortality (Percentage of Participants Who Died Due to Causes Other Than Study Cancer)
Description: Failure is defined as Death from second primary, protocol treatment, or "other cause". Failure time is defined as time from randomization to first occurrence of failure, death due to study cancer or unknown cause (competing risk), or last follow-up (censored). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year estimates are provided.
Time Frame: as for outcome 2
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT+ Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 63 | 123
percentage of participants | 5.3 [1.4 to 13.4] | 10.5 [5.7 to 17.0]
Statistical Analysis 1: Comparison: RT+ Cetuximab vs RT + Durvalumab; Test type: Superiority; p = 0.3201, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.75, 95% CI 2-sided [0.57 to 5.38]

7. Secondary Outcome: Percentage of Participants With Complete or Partial Response at 4-month Scan Determined by Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1
Description: Fludeoxyglucose F-18 positron emission tomography/computed tomography (FDG-PET/CT) scans at baseline and four months after the end of radiation therapy are compared.
  Per RECIST 1.1:
  * Complete response:
    * Disappearance of all lesions and pathologic lymph nodes
  * Partial response:
    * ≥ 30% decrease sum of the longest diameters
    * No new lesions
    * No progression of non-target lesions
Time Frame: Baseline and 4 months after end of RT (approximately 6.5 months)
Population: Randomized participants with 4-month response assessed by PET
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT+ Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 22 | 29
percentage of participants | 72.7 [51.8 to 86.8] | 75.9 [57.9 to 87.8]
Statistical Analysis 1: Comparison: RT+ Cetuximab vs RT + Durvalumab; Test type: Superiority; p = 1.00, Fisher Exact — Two-sided significance level = 0.05

8. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 5.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to last follow-up: weekly during RT, RT end, from end of RT: months 1, (Cetuximab: 2, 3,) 4, 8, 12, 18, 24, 30, 36, then annually. Additionally, prior to each adjuvant durvalumab cycle. Maximum follow-up at time of analysis= 4.2 yr.
Population: Randomized and started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RT+ Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 61 | 119
Participants
  < Grade 3 | 12 | 36
  Grade 3 | 37 | 57
  Grade 4 | 11 | 15
  Grade 5 | 1 | 11
Statistical Analysis 1: Comparison: RT+ Cetuximab vs RT + Durvalumab; Test type: Superiority; p = 0.0688, Fisher Exact — Two-side significance level = 0.05

9. Secondary Outcome: Change in Quality of Life (QOL) Analysis
Description: Assessed using European Organization for Research and Treatment of Cancer Core Questionnaire (EORTC QLQ)/Head-and-Neck module (H&N35), EuroQol- 5 Dimension (EQ5D), M. D. Anderson Dysphagia Inventory (MDADI), patient reported outcomes (PRO)-CTCAE, geriatric screening (G8). The mean summary score of the EORTC QLQ/H&N35, EQ5D, MDADI, PRO-CTCAE, G8, CCI, and the subscales will be determined. The mean change from baseline at each time point will be summarized using mean and standard deviations for each arm. Mean change from baseline will be compared between the arms using a two sample t test. If data normality assumptions are not met, the Wilcoxon rank sum test will be used to test the hypothesis. Mean change from baseline will be tested using an omnibus F test followed by individual comparisons of change scores at different time points within each treatment group. The same analysis will be conducted for between group comparisons at each time point.
Time Frame: Baseline up to 12 months
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Change in Swallowing QOL Using Total Composite M. D. Anderson Dysphagia Inventory (MDADI) Score
Description: The mean change from baseline at each time point will be summarized using mean and standard deviations for each arm. Mean change from baseline will be compared between the arms using a two sample t test. If data normality assumptions are not met, the Wilcoxon rank sum test will be used to test the hypothesis.
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted, anticipated posting 2026-06

11. Secondary Outcome: Progression-free Survival (Percentage of Participants Alive Without Progression) by Baseline PD-L1 (Programmed Cell Death Ligand 1) Expression
Description: Failure for progression-free survival is defined as local, regional, or distant disease progression, or death from any cause. Progression was assessed by imaging, clinical assessment, or biopsy. Failure time is defined as time from randomization to failure or last follow-up (censored). PD-L1 expression is defined by a combined positive score (CPS) ≥ 1, assessed by masked central analysis of baseline tissue specimens. CPS = [(number of tumor cells positive for PD-L1) / (number of tumor cells positive for PD-L1 + number of tumor cells negative for PD-L1)] multiplied by 100, yielding a possible score of 0 to 100. Treatment effect hazard ratios within PD-L1 subgroup were estimated by Cox proportional hazards model and progression-free survival estimates were estimated by Kaplan-Meier method. Analysis was planned to occur after 69 failure events had been reported and tissue specimen analysis was complete.
Time Frame: From randomization to date of progression or last follow-up, whichever occurs first. Maximum follow-up at time of analysis was 4.2 years. Two-year PFS estimates are reported.
Population: Randomized participants with CPS score.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 52 | 108
percentage of participants
  CPS ≥ 1 (PD-L1 expression): number analyzed (Participants) | 39 | 88
  CPS ≥ 1 (PD-L1 expression) | 59.9 [43.6 to 76.2] | 54.8 [43.9 to 65.6]
  CPS = 0 (no PD-L1 expression): number analyzed (Participants) | 13 | 20
  CPS = 0 (no PD-L1 expression) | 61.5 [35.1 to 88.0] | 30.0 [9.9 to 50.1]
Statistical Analysis 1: Comparison: RT + Cetuximab vs RT + Durvalumab; CPS ≥ 1; Test type: Superiority; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.62 to 1.97] — Reference arm = RT + Cetuximab
Statistical Analysis 2: Comparison: RT + Cetuximab vs RT + Durvalumab; CPS = 0; Test type: Superiority; Cox Proportional Hazard = 1.64, 95% CI 2-sided [0.66 to 4.06] — Reference arm = RT + Cetuximab
Statistical Analysis 3: Comparison: RT + Cetuximab vs RT + Durvalumab; Interaction; Test type: Superiority; p = 0.41, Regression, Cox — Testing the interaction of treatment arm and PD-L1 expression (CPS ≥ 1, CPS = 0)

12. Secondary Outcome: Progression-free Survival (Percentage of Participants Alive Without Progression) by Baseline p16 Status
Description: Failure for progression-free survival is defined as local, regional, or distant disease progression, or death from any cause. Progression was assessed by imaging, clinical assessment, or biopsy. Failure time is defined as time from randomization to failure or last follow-up (censored). Positive p16 status was defined as more than 70% strong nuclear or nuclear and cytoplasmic staining of tumor cells, confirmed by central pathology review. Treatment effect hazard ratios within p16 subgroup were estimated by Cox proportional hazards model and progression-free survival estimates were estimated by Kaplan-Meier method. Analysis was planned to occur after 69 failure events had been reported and tissue specimen analysis was complete.
Time Frame: as for outcome 11
Population: Randomized participants with p16 status.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RT + Cetuximab | RT + Durvalumab
Number analyzed (Participants) | 59 | 115
percentage of participants
  p16-positive: number analyzed (Participants) | 33 | 68
  p16-positive | 74.8 [59.6 to 89.9] | 68.8 [57.4 to 80.1]
  p16-negative: number analyzed (Participants) | 26 | 47
  p16-negative | 48.1 [27.6 to 68.5] | 23.2 [10.1 to 36.3]
Statistical Analysis 1: Comparison: RT + Cetuximab vs RT + Durvalumab; p16-positive; Test type: Superiority; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.57 to 2.51] — Reference arm = RT + cetuximab
Statistical Analysis 2: Comparison: RT + Cetuximab vs RT + Durvalumab; p16-negative; Test type: Superiority; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.83 to 2.89] — Reference arm = RT + cetuximab
Statistical Analysis 3: Comparison: RT + Cetuximab vs RT + Durvalumab; Interaction; Test type: Superiority; p = 0.61, Regression, Cox — Testing the interaction of treatment arm and p16 status (positive, negative)

13. Other Pre Specified Outcome: Secondary Biomarker Analysis
Description: Will perform multiparametric flow cytometry on peripheral mononuclear cells (PBMC) from patient-derived blood samples to quantify changes in immune cell frequency and activation status before, during and after radiation combined with cetuximab or radiation combined with durvalumab. To assess the statistical significance of pre- to post-treatment changes in levels of immunoglobulin (Ig)Gs as well as other markers, normalized signal intensities (log2) will be tested using a paired t test within an arm and two sample t test between the two arms. If the distribution assumption is violated for the t tests, nonparametric tests, such as the Wilcoxon signed-rank test will be considered. Lastly, the association between PFS and OS and post-treatment changes in frequency and activation state of T-cells, clonality and diversity of T cell receptor (TCR), and IgG levels will be evaluated using a two-sided Wald test at 0.05 level on the basis of Cox models.
Time Frame: Baseline up to 4 months after RT
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: PRO-CTCAE is not intended for expedited reporting, real time review or safety reporting. PRO-CTCAE data are exploratory and not currently intended for use in data safety monitoring or adverse event stopping rules.
Time Frame: Up to 3 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: QOL Endpoints Using Other Items in EORTC QLQ/HN35, EQ5D and MDADI Subscales
Description: The mean change from baseline at each time point will be summarized using mean and standard deviations for each arm. Mean change from baseline will be compared between the arms using a two sample t test. If data normality assumptions are not met, the Wilcoxon rank sum test will be used to test the hypothesis. Mean change from baseline will be tested using an omnibus F test followed by individual comparisons of change scores at different time points within each treatment group. The same analysis will be conducted for between group comparisons at each time point.
Time Frame: Up to 12-24 months from end of RT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Weekly during RT, RT end, from end of RT: months 1, (Cetuximab: 2, 3,) 4, 8, 12, 18, 24, 30, 36, then annually. Additionally, prior to each adjuvant durvalumab cycle. Maximum follow-up at time of analysis= 4.2 yr.
Description: All-cause mortality was assessed in all enrolled participants. Adverse events were assessed in enrolled participants who started study treatment. CTCAE 4.0 was used in the lead-in component and CTCAE 5.0 was used in the phase II component.
Arm/Group | (Lead-in) RT + Durvalumab | RT + Cetuximab | RT + Durvalumab
All-Cause Mortality (participants affected / at risk) | 3/10 | 17/63 | 41/123
Serious Adverse Events (participants affected / at risk) | 4/10 | 51/61 | 84/119
Other Adverse Events (participants affected / at risk) | 10/10 | 61/61 | 118/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Lead-in) RT + Durvalumab (N=10) | RT + Cetuximab (N=61) | RT + Durvalumab (N=119)
Anemia (Blood and lymphatic system disorders) | 0 | 5 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 1
Heart failure (Cardiac disorders) | 0 | 3 | 3
Myocardial infarction (Cardiac disorders) | 0 | 1 | 5
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Vision decreased (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Anal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 18 | 25
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 2 | 1
Ileal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 11 | 14
Nausea (Gastrointestinal disorders) | 0 | 2 | 4
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Oral pain (Gastrointestinal disorders) | 0 | 3 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Chills (General disorders) | 0 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 3
Edema limbs (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 8
Fever (General disorders) | 0 | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Sudden death NOS (General disorders) | 0 | 1 | 4
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 1 | 0
Bone infection (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 4 | 5
Sepsis (Infections and infestations) | 0 | 1 | 2
Skin infection (Infections and infestations) | 0 | 1 | 3
Stoma site infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 8 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4
Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1 | 3
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 2
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 19 | 30
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Serum amylase increased (Investigations) | 0 | 0 | 2
Weight loss (Investigations) | 0 | 5 | 11
White blood cell decreased (Investigations) | 0 | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 7 | 17
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 6
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 3
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 2
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 5
Hypotension (Vascular disorders) | 0 | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (Lead-in) RT + Durvalumab (N=10) | RT + Cetuximab (N=61) | RT + Durvalumab (N=119)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 19 | 43
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 2 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 2
Conduction disorder (Cardiac disorders) | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 6
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 7 | 13
Hearing impaired (Ear and labyrinth disorders) | 0 | 3 | 6
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 13
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Endocrine disorders - Other (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 10
Hypothyroidism (Endocrine disorders) | 4 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 7 | 25
Blurred vision (Eye disorders) | 0 | 0 | 3
Dry eye (Eye disorders) | 0 | 1 | 1
Eye disorders - Other (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Papilledema (Eye disorders) | 0 | 0 | 1
Vision decreased (Eye disorders) | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 12 | 17
Anal pain (Gastrointestinal disorders) | 0 | 1 | 1
Belching (Gastrointestinal disorders) | 0 | 1 | 2
Bloating (Gastrointestinal disorders) | 0 | 0 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 25 | 40
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 17 | 31
Dry mouth (Gastrointestinal disorders) | 10 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 37 | 84
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 3
Dysphagia (Gastrointestinal disorders) | 9 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 47 | 97
Esophageal pain (Gastrointestinal disorders) | 0 | 2 | 2
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 7
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 7 | 6
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 7 | 15
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 7 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 46 | 85
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 35 | 52
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 10 | 6
Rectal pain (Gastrointestinal disorders) | 0 | 2 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 5 | 6
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 19 | 24
Chills (General disorders) | 0 | 2 | 5
Edema face (General disorders) | 0 | 3 | 7
Edema limbs (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 14 | 29
Fatigue (General disorders) | 7 | 0 | 0
Fatigue (General disorders) | 0 | 52 | 98
Fever (General disorders) | 0 | 3 | 7
Gait disturbance (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
General disorders and administration site conditions - Other (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 6 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1
Localized edema (General disorders) | 0 | 1 | 5
Malaise (General disorders) | 0 | 0 | 1
Neck edema (General disorders) | 4 | 0 | 0
Neck edema (General disorders) | 0 | 2 | 8
Non-cardiac chest pain (General disorders) | 0 | 1 | 3
Pain (General disorders) | 3 | 0 | 0
Pain (General disorders) | 0 | 8 | 20
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 1
Bone infection (Infections and infestations) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Esophageal infection (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 2 | 6
Laryngitis (Infections and infestations) | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 2 | 8
Mucosal infection (Infections and infestations) | 0 | 2 | 1
Myelitis (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 0 | 3
Paronychia (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Shingles (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 3
Skin infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 2 | 7
Thrush (Infections and infestations) | 0 | 6 | 14
Tooth infection (Infections and infestations) | 0 | 1 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 9 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 44 | 83
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 8
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 0 | 3
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 6 | 14
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 4 | 12
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 9 | 20
Blood bicarbonate decreased (Investigations) | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1
CPK increased (Investigations) | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 2 | 4
Cardiac troponin T increased (Investigations) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 11 | 25
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 6
Investigations - Other (Investigations) | 0 | 2 | 5
Lipase increased (Investigations) | 0 | 0 | 9
Lymphocyte count decreased (Investigations) | 4 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 28 | 47
Neutrophil count decreased (Investigations) | 0 | 2 | 4
Platelet count decreased (Investigations) | 0 | 5 | 16
Serum amylase increased (Investigations) | 0 | 0 | 8
Thyroid stimulating hormone increased (Investigations) | 0 | 4 | 4
Weight gain (Investigations) | 0 | 2 | 3
Weight loss (Investigations) | 8 | 0 | 0
Weight loss (Investigations) | 0 | 32 | 67
White blood cell decreased (Investigations) | 0 | 8 | 15
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 6 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 31 | 67
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 13 | 25
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 14 | 30
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 4 | 6
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypernatremia (Metabolism and nutrition disorders) | 0 | 4 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 16 | 22
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 7 | 15
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 7 | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 20 | 21
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 9 | 28
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 9 | 25
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 8 | 16
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 1
Aphonia (Nervous system disorders) | 0 | 0 | 1
Brachial plexopathy (Nervous system disorders) | 0 | 1 | 1
Concentration impairment (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 23
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 6 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 35 | 73
Dysphasia (Nervous system disorders) | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 13 | 12
Lethargy (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Meningismus (Nervous system disorders) | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 5 | 12
Presyncope (Nervous system disorders) | 0 | 0 | 3
Radiculitis (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 2
Stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 5 | 10
Confusion (Psychiatric disorders) | 0 | 1 | 2
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 4 | 8
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 9 | 11
Psychiatric disorders - Other (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 5
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Glucosuria (Renal and urinary disorders) | 0 | 0 | 3
Hematuria (Renal and urinary disorders) | 0 | 1 | 3
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 3
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 2 | 2
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 3 | 6
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 2
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 28 | 54
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 42
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 14 | 18
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 7
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 11
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 23 | 38
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 13
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 8 | 13
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 23 | 31
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 41 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 14 | 24
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 7 | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 2 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 14 | 17
Hypotension (Vascular disorders) | 0 | 8 | 14
Lymphedema (Vascular disorders) | 3 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 13 | 17
Thromboembolic event (Vascular disorders) | 0 | 2 | 1
Vascular disorders - Other (Vascular disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Phase II (phII) component stopped enrollment early due to toxicity and futility concerns, with 186 of the 234 planned participants, but continued to collect data required for the final phII analysis. Per the protocol, the study did not continue to phase III (phIII). Therefore, the phIII primary outcome measure (OM) of overall survival was analyzed as a phII secondary OM. Accordingly, the phIII PD-L1 and p16 analyses were analyzed using the phII primary OM of progression-free survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval from the sponsor. In addition, PI's are required to abide by Collaborator's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03258554/Prot_SAP_000.pdf